CLINICAL TRIAL: NCT06469658
Title: Personalized Management of Type 2 Diabetes Using AI-Guided (GenAIS TM) Dietary Supplementation: A Randomized Controlled Clinical Trial
Brief Title: Personalized Management of Type 2 Diabetes Using AI-Guided (GenAIS TM) Dietary Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Triangel Scientific (Industry); Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW014
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Diabetes
Keywords: AI-guided dietary supplementation; Personalized supplementation; HbA1c reduction; Genetic and metabolic profiling
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Other: The standard practice dietary supplements intervention
- Group 2 (Experimental)
  Interventions: Other: The AI-guided practice dietary supplements group

INTERVENTIONS:
Other: The standard practice dietary supplements intervention — Participants receive supplements prescriptions from a physician based on current standard practices, which include biochemical markers, genetic data, and metabolic profiles.
  Arms: Group 1
Other: The AI-guided practice dietary supplements group — Participants receive DS prescriptions determined by GenAIS, an AI system which considers genetic data, metabolic profiles, biochemical markers, and patient history.
  Arms: Group 2

SUMMARY:
This randomized controlled trial investigates the effectiveness of AI-guided dietary supplement prescriptions compared to standard physician-guided prescriptions in managing Type 2 diabetes (T2D). The study includes 160 participants with T2D, aged 40-75, who will be randomly assigned to either the control group (standard physician-guided prescriptions) or the AI-guided group (prescriptions determined by GenAIS, an AI system by Triangel Scientific). The primary objective is to compare the reduction in HbA1c levels between the two groups over 6 months. Secondary outcomes include changes in fasting glucose, lipid profiles, body weight, BMI, hsCRP levels, and adherence to the dietary supplement regimen. The AI system integrates genetic, metabolic, and clinical data to provide personalized supplement recommendations, aiming to improve glycemic control and overall metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75 years.
* Diagnosed with Type 2 diabetes (HbA1c between 7.0% and 10.0%).
* Stable anti-diabetic medication regimen for at least 3 months prior to the study.
* Willingness to provide genetic and metabolic data.

Exclusion Criteria:

* Type 1 diabetes or other specific types of diabetes.
* Significant renal, hepatic, or cardiovascular diseases.
* Use of dietary supplements that affect glucose metabolism within the last 3 months.
* Pregnancy or breastfeeding

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c levels | 180 days

SECONDARY OUTCOMES:
Percent change in fasting venous blood glucose levels. | 180 days
Percent change in high-sensitivity C-reactive protein | 180 days
Percent change in cholesterol | 180 days
Percent change in HDL-C, | 180 days
Percent change in LDL-C | 180 days
Percent change in triglycerides | 180 days
Percent change in body weight | 180 days
Incidence of any adverse effects related to supplements | 180 days
Percent change in Body mass index (BMI) | 180 days
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | 180 days
fasting insulin levels change (mU/mL) | 180 days
Waist Circumference (cm) change | 180 days
microalbuminuria (%) difference | 180 days
changes in physical activity levels (hours/week) | 180 days
Percentage of participants using antihypertensive medications (%) | 180 days
Percentage of participants using antihypertensive medications (%). | 180 days
Percentage of participants using lipid-lowering medications (%). | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia